All statistical analyses were conducted using InStat 3.1a (GraphPad Software, La Jolla, CA). A modified intent-to-treat (ITT) population was used for analyses. For each outcome variable, the modified ITT population included all subjects with at least one post-baseline psychometric measurement (subjects received at least one week of aripiprazole). Demographic data is presented as means and standard deviations while bivariant data were contrasted using paired-t tests. A repeated measure analysis of variance (ANOVA) model was used to assess the changes in the psychometric tests. In cases where a subject did not complete the entire 6-week trial, the last available observation was carried forward (LOCF) and used for statistical comparisons. A repeated measure analysis of variance was used to assess the changes in the psychometric tests. For determining significance of statistical tests  $\langle$  was set at 0.05.